CLINICAL TRIAL: NCT04085965
Title: Testing the Feasibility and Preliminary Effect of Summer Day Camp on Excess Summer Weight Gain in Children From Low-income Communities
Brief Title: Testing the Feasibility and Preliminary Effect of Summer Camp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Hassenfeld Child Health Innovation Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 710-9073
Record Dates: First submitted 2019-09-03; First posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Childhood Obesity Prevention
Keywords: Summer Camp; Child overweight / obesity; Diet; Physical Activity
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAMP (Experimental): Children randomized to CAMP were enrolled in the Boys and Girls Club Camp in one of two low-income Rhode Island communities in summer 2017 or 2018 for 7-weeks in 2017 and 8-weeks in 2018 due to a delayed end to the 2017 school year (i.e. snow days). Camp was offered daily from 8:30 to 4:30.
  Interventions: Behavioral: Boys and Girls Club summer day camp
- Summer As Usual (No Intervention): Children randomized to the SAU group were asked to experience an unstructured summer as otherwise planned by their parent / guardian. They agreed to not attend structured summer programming (i.e. camp, summer school, or day care) for more than one week over the summer so as to provide an inactive control group for comparison to those in CAMP.

INTERVENTIONS:
Behavioral: Boys and Girls Club summer day camp — Daily camp activities included sports, games, obstacle courses, swimming and boating, summer learning and arts and crafts. Lunch was served daily via the USDA's Summer Food Service Program.
  Arms: CAMP

SUMMARY:
This pilot randomized controlled trial was designed to assess the feasibility and preliminary efficacy of randomizing children, ages 6-12 years from two low-income communities in Rhode Island, to attend a summer day camp (CAMP) or to experience summer as usual (SAU). Children randomized to CAMP attended a Boys and Girls Club summer day camp for 8-weeks in summer 2017 or 2018. As part of the consent process, children randomized to SAU agreed to experience an unstructured summer (i.e. not enroll in more than one week of summer camp, summer school or other structured summer programming). Primary feasibility outcomes included retention, engagement and completion of midsummer measures. Secondary outcomes, change in BMIz (a proxy for excess summer weight gain), physical activity engagement, sedentary behavior, and diet (energy intake and diet quality), were collected by blinded research staff at the end of the school year, midsummer and the end of the summer.

ELIGIBILITY:
Inclusion Criteria:

* Qualify for free or reduced-price meals at school
* Speak English (for purposes of camp participation)
* Agree, along with their parent(s), to randomization.

Exclusion Criteria:

* A medical condition that interferes with participation in physical activity
* Enrollment in summer programming (camp, summer school, etc) for more than one week

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Retention | Baseline to end of summer; 8 weeks
  Number of participants who completed both baseline and end of summer assessments
Camp Attendance | 8 weeks
  Number of days children attended the Boys and Girls Club Camp
Participation in Summer Activities | 8 weeks
  Number of days children attended camp, summer school, or day care over the summer
Completion of study measures | Baseline (May / June); Midsummer (mid-July)
  Number of participants who completed three 24-hour diet recalls and/or 7-days of actigraphy at baseline and mid-summer assessment visits

SECONDARY OUTCOMES:
Excess summer weight gain | Baseline to end of summer; 8 weeks
  Change in BMIz
Physical Activity | 4-6 weeks (from baseline (end of May / beginning of June) to mid-summer (mid-July))
  Change in minutes of moderate to vigorous physical activity (MVPA) as measured by ActiGraph accelerometer
Sedentary Behavior | 4-6 weeks (from baseline (end of May / beginning of June) to mid-summer (mid-July))
  Change in percent time spent sedentary as measured by ActiGraph accelerometer
Energy Intake | 4-6 weeks (from baseline (end of May / beginning of June) to mid-summer (mid-July))
  Change in total energy intake as measured from 3 non-consecutive 24-hour diet recalls
Diet Quality | 4-6 weeks (from baseline (end of May / beginning of June) to mid-summer (mid-July))
  Change in Diet Quality as measured by the HEI-2015 from three non-consecutive 24-hour diet recalls

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evans EW, Wing RR, Pierre DF, Howie WC, Brinker M, Jelalian E. Testing the effect of summer camp on excess summer weight gain in youth from low-income households: a randomized controlled trial. BMC Public Health. 2020 Nov 17;20(1):1732. doi: 10.1186/s12889-020-09806-y. PMID 33203385